CLINICAL TRIAL: NCT01638650
Title: To Determine the Effect of the Modified SQV/r (Saquinavir-boosted by Ritonavir) Regimen (500/100 mg for the 1st Week Followed by 1000/100 mg for the 2nd Week) on the QTc Interval, Pharmacokinetics, and Antiviral Activity in Treatment-naive HIV-1 Infected Patients
Brief Title: A Study of Ritonavir-Boosted Invirase (Saquinavir) in Treatment-Naïve HIV-1 Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25607
Record Dates: First submitted 2012-06-06; First posted 2012-07-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Saquinavir

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTIs); Drug: ritonavir; Drug: saquinavir [Invirase]

INTERVENTIONS:
Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTIs) — in accordance with current clinical HIV treatment guidelines
Drug: ritonavir — 100 mg bid orally, Days 1-14
Drug: saquinavir [Invirase] — 500 mg bid orally Days 1-7, 1000 mg bid orally Days 8-14

SUMMARY:
This open-label study will evaluate the safety, pharmacokinetics and antiviral activity of a modified Invirase (saquinavir)/ritonavir regimen in treatment-naïve HIV-1 infected patients. Patients will receive Invirase 500 mg plus ritonavir 100 mg twice daily orally for the first week, followed by Invirase 1000 mg plus ritonavir 100 mg twice daily orally for the second week. The study treatment will be given in combination with two Nucleoside Reverse Transcriptase Inhibitors (NRTIs), in accordance with the current clinical HIV treatment guidelines. Anticipated time on study treatment is 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* HIV-1 infection
* Currently treatment-naïve and eligible to initiate a ritonavir-boosted Protease Inhibitor based regimen and willing and able to initiate saquinavir/ritonavir therapy for the first 14 days; the saquinavir/ritonavir regimen will be in combination with two Nucleoside Reverse Transcriptase Inhibitors (NRTIs), in accordance with the current clinical HIV treatment guidelines
* Body mass index 18-32 kg/m2, inclusive
* Female patients of childbearing potential and male patients with female partners of childbearing potential must use 2 methods of contraception as defined by protocol during the study and for at least one month after the last dose of study drug
* Non-smoker or patients who have stopped smoking more than three months prior to Day 1 of the study

Exclusion Criteria:

* Coinfection with hepatitis B or C (acute or chronic)
* Anticipated use or need for significant concomitant medical treatment during the study period, other than background antiretroviral therapy
* Participation in a clinical study with an investigational drug or device within 3 months prior to Day 1 of the study
* Pregnant or lactating women
* Any clinically relevant history of substance abuse or addiction including alcohol and/or other drugs of abuse
* Special dietary restrictions that would prohibit consumption of standardized meal (e.g. vegetarian, vegan, gluten-free, lactose-free, kosher)
* Decompensated liver disease
* Congenital or documented acquired QT prolongation
* Electrolyte disturbances, particularly uncorrected hypokalaemia
* Clinically relevant bradycardia
* Clinically relevant heart failure with reduced left-ventricular ejection fraction
* Previous history of symptomatic arrhythmias
* History of clinically significant gastro-intestinal, renal, hepatic, bronchopulmonary, neurological, psychiatric, cardiovascular, endocrinological, , hematological, or allergic disease, metabolic disorder, cancer, or cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Maximal increase in QTc interval (continuous Holter 12-lead ECG monitoring time points Days 1, 3, 4, 7, 10 and 14) | 14 days

SECONDARY OUTCOMES:
Pharmacokinetics: Plasma concentrations | Pre-dose and 2, 4, 6, 8 and 12 hours post-dose, Days 3, 4, 7, 10 and 14
Pharmacodynamics: Change in HIV-RNA levels | from baseline to Day 14
Safety: Incidence of adverse events | approximately 6 months
Change in ECG parameters | from baseline to Day 14
Correlation between saquinavir plasma concentration and QTc interval changes | approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- London, United Kingdom